CLINICAL TRIAL: NCT06533852
Title: Fecal Microbiome Transplantation in Cirrhosis: Randomized, Double-blinded, Placebo-Controlled Trial in Patients With Decompensated Cirrhosis
Brief Title: Fecal Microbiome Transplantation in Cirrhosis: Trial in Patients With Decompensated Cirrhosis
Acronym: LiverGut
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-509151-13-00
Record Dates: First submitted 2024-07-15; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal Microbiome Transplantation (FMT) (Experimental): A first dose of 24 capsules of FMT at baseline and a second dose of 24 capsules of FMT at 3 months. Each dose (24 capsules) contains approximately 50g of stool.
  Interventions: Drug: Fecal Microbiome Transplantation (FMT)
- FMT Placebo (Placebo Comparator): A first dose of 24 capsules of FMT placebo at baseline and a second dose of 24 capsules of FMT placebo at 3 months. Each dose (24 capsules) contains in total 6 g of microcrystalline cellulose or equivalent.
  Interventions: Other: FMT Placebo

INTERVENTIONS:
Drug: Fecal Microbiome Transplantation (FMT) — Two doses:
  First dose: 24 capsules of FMT at baseline. Second dose: 24 capsules of FMT at 3 months.
  Arms: Fecal Microbiome Transplantation (FMT)
Other: FMT Placebo — Two doses:
  First dose: 24 capsules of FMT placebo at baseline. Second dose: 24 capsules of FMT placebo at 3 months.
  Arms: FMT Placebo

SUMMARY:
This is a phase III, multicenter, double-blind, placebo-controlled, randomized clinical trial to evaluate the safety and efficacy of Fecal Microbiota Transplantation (FMT) from healthy subjects to patients with decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Cirrhosis defined by standard clinical criteria, ultrasonographic findings and/or histology. Cirrhosis of any etiology may be included except from patients with cirrhosis due to autoimmune hepatitis, and patients with cirrhosis due to cholestatic liver disease can only be included in the study if they present clinical decompensation of cirrhosis (i.e. ascites).
3. Child-Pugh B or C patients (7- up to 12 points).
4. Women of child-bearing potential* must have a negative pregnancy test in serum before the inclusion in the study and agree to use highly effective contraceptive methods during the study. Highly effective contraceptive methods will include: intrauterine device, bilateral tubal occlusion, vasectomized partner and sexual abstinence** (only if refraining from heterosexual intercourse during the period of twelve months). Hormonal contraceptive methods will be avoided due to the risk of adverse events and impairment of liver function.

Exclusion Criteria:

1. Previous history of gastrointestinal surgery or colorectal cancer.
2. Patients with previous history of intestinal obstruction or those who are at increased risk of this complication.
3. Active Clostridium Difficile infection.
4. Patients on treatment with non-selective beta-blockers for <3 month or without stable doses.
5. Patients on treatment with any immunosuppressive drugs.
6. Patients on antiviral therapy for HCV or those who have received it within the last 12 months.
7. Patients on antiviral therapy for HBV therapy for < 12 months.
8. Patients with hepatocellular carcinoma, except for patients with early HCC (BCLC-0 or BCLC-A) or patients with previous history of HCC and absence of recurrence 2 years after treatment.
9. Patients admitted to the hospital for acute decompensation of the disease. These patients could be included after discharged as long as they do not present any of the following events:

   1. Bacterial infection within 10 days before study inclusion.
   2. Gastrointestinal bleeding within 10 days before study inclusion.
   3. Current overt hepatic encephalopathy, defined as grade II-IV hepatic encephalopathy according to the New-Haven classification.
10. Patients with ACLF according to the criteria published by Moreau et al. (Appendix 1).
11. Severe alcoholic hepatitis requiring corticosteroid therapy (MELD > 20) in the last 6 months.
12. Patients with active alcohol consumption of more than 21 units per week.
13. HIV infection.
14. Patients with a history of significant extra hepatic disease with impaired short-term prognosis, including congestive heart failure New York Heart Association Grade III/IV, COPD GOLD >2, chronic kidney disease with serum creatinine >2mg/dL or under renal replacement therapy.
15. Patients with current extra hepatic malignancies including solid tumours and hematologic disorders.
16. Patients with previous organ transplantation.
17. Pregnancy or breastfeeding.
18. Patients included in other clinical trials in the month before inclusion.
19. Patients with mental incapacity, language barrier, bad social support or any other reason considered by the investigator precluding adequate understanding, cooperation or compliance in the study.
20. Refusal to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment in halting the progression of decompensated cirrhosis. | Screening to month 12.
  Assessed by time to first decompensation event (acute kidney injury (AKI), ascites, bacterial infection, gastrointestinal bleeding, HE).

SECONDARY OUTCOMES:
Time to transplant-free survival | At month 1, month 3, month 6 and month 12
  Assessed by transplant-free survival
Mortality rates | At month 1, month 3, month 6 and month 12
  Assessed by mortality rates
Rate of patients developing/ worsening individual complications of cirrhosis. | At baseline, month 1, month 3, month 6 and month 12.
  Assessed by ascites, acute kidney injury, bacterial infections, gastrointestinal bleeding and hepatic encephalopathy.
Frequency of hospital admissions due to complications of cirrhosis. | At baseline, 1 month, 3 months, 6 months and 12 months.
  Assessed by hospital admissions due to complications of cirrhosis.
Development of acute-on-chronic liver failure (ACLF) | At baseline, 1 month, 3 months, 6 months and 12 months.
  Assessed by time to first episode of ACLF
Development of acute-on-chronic liver failure (ACLF) | At month 3, month 6 and month 12.
  Assessed by total number of patients developing ACLF
Development of acute-on-chronic liver failure (ACLF) | At baseline, 1 month, 3 months, 6 months and 12 months.
  Assessed by severity of ACLF episodes based on ACLF grade (from grade 1 to grade 3) and CLIF-C-ACLF score
Development of acute-on-chronic liver failure (ACLF) | At baseline, 1 month, 3 months, 6 months and 12 months.
  Assessed by number and type of organ failures
Changes from baseline in systemic inflammatory response. | At baseline, 1 month, 3 months, 6 months and 12 months.
  Evaluated by measurement in a large array of plasma cytokine levels including, but not limited to TNFα, IL-6, IL8, IL-10, IL-1β, IFN-ɣ, G-CSF, VCAM, VEGF, as well as an oxidized form of albumin, human nonmercaptalbumin-2 (HNA2).
PBMCs phenotype and function. | At baseline, 1 month, 3 months, 6 months and 12 months.
  Analysed by flow cytometry, functional analysis, and RNAseq single cell analysis.
Changes from baseline in different plasma and urine prognostic biomarkers. | At baseline, 1 month, 3 months, 6 months, and 12 months.
  Measurated by different plasma and urine prognostic biomarkers including, but not only, copeptin, NGAL, PD-L1, L-FABP.
Changes from baseline in systemic hemodynamics and vasoactive hormones. | At baseline, 1 month, 3 months, 6 months and 12 months.
  Measurated by systemic hemodynamics and vasoactive hormones: plasma renin concentration and plasma copeptin.
Changes from baseline in blood levels of bacterial DNA or bacterial products. | At baseline, 1 month, 3 months, 6 months and 12 months.
  Measurated by blood levels of bacterial DNA or bacterial products.
Changes from baseline in liver function. | At baseline, 1 month, 3 months, 6 months and 12 months.
  Evaluated by MELD (Model for End-stage Liver Disease) score.
Changes from baseline in liver function. | At baseline, 1 month, 3 months, 6 months and 12 months.
  Evaluated by CLIF-AD score.
Changes from baseline in liver function. | At baseline, 1 month, 3 months, 6 months and 12 months.
  Evaluated by Child Pugh Score.(from 1 point to 15 points)
Analyze microbiome composition from saliva and stool. | At baseline, and months 1, 3 and 6.
  Measurated by analysis of microbial genes.
Changes in hepatic venous pressure gradient (HVPG) from baseline. | At baseline and month 6.
  Measurated by the hepatic venous pressure gradient.
Assess Quality of life, functional assessment and in Minimal Hepatic Encephalopathy. | At baseline, 3 months, 6 months and 12 months.
  Evaluated with data obtained from CLDQ (Chronic Liver Disease Questionnaire) questionnaire.
Assess Quality of life, functional assessment and in Minimal Hepatic Encephalopathy. | At baseline, 3 months, 6 months and 12 months.
  Evaluated with data obtained from Liver Frailty Index.
Assess Quality of life, functional assessment and in Minimal Hepatic Encephalopathy. | At baseline, 3 months, 6 months and 12 months.
  Evaluated with data obtained from PHES (Psychometric Hepatic Encephalopathy Score) questionnaire.
Changes from baseline in AUDIT test. | AUDIT test at baseline, 3 months, 6 months and 12 months
  Evaluated from AUDIT test
Changes from baseline in alcohol consumption. | PETh measurament test at baseline, 1 month, 3 months, 6 months and 12 months.
  Evaluated from PETh measurament.
Assess the effect of FMT in ECG (Electrocardiogram). | At screening, baseline and months 3,6 and 12.
  Evaluated by changes in ACE score.
Proportion of patients with treatment-related adverse events. | Screening to month 12.
  Evaluated by treatment-related adverse events.
Proportion of patients with severe treatment-related adverse events. | Screening to month 12.
  Evaluated by treatment-related adverse events.